CLINICAL TRIAL: NCT02273830
Title: Benefits of Liquid Oxygen in COPD Patients Presenting Desaturation on Exercise But Without Conventional Criteria for Domiciliary Oxygen Therapy.
Brief Title: Benefits of Liquid Oxygen in COPD Patients Presenting Desaturation During Exercise.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jtarrega (Other)
Collaborators: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other); Hospital Mutua de Terrassa (Other); Hospital Dos de Maig (Unknown); Hospital Universitari Sant Joan de Reus (Other)
Responsible Party: Sponsor-Investigator, Jtarrega, PhD, Hospital de Granollers
Organization: Hospital de Granollers (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 20131001
Record Dates: First submitted 2014-10-22; First posted 2014-10-24 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: oxygen therapy; COPD; exercise
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity | interventions — Oxygen

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- oxygen adjusted (Active Comparator): oxygen adjusted to get SpO2> 90% during the walking test
  Interventions: Drug: oxygen
- control group (Placebo Comparator): oxygen at 3L/min
  Interventions: Drug: oxygen

INTERVENTIONS:
Drug: oxygen — Oxygen administered after adjustment during a waking test or at 3L/min

SUMMARY:
The purpose of this study is analyzed the impact of oxygen adjusted during exercise in COPD patients without conventional for LTOT but with exercise desaturation.

DETAILED DESCRIPTION:
Oxygen will be administered through nasal cannulae. Patients will be provided with a tank of liquid oxygen and a rechargeable portable device. The 6 minuts walking test will be used to adjusted oxygen flow in the GFA group (to achieve a mean SpO2 ≥ 90%). In the control group (GC), a 3L/min oxygen flow will be administer. Oxygen is used when the patient perform physical activity. The treatment period for each patient is 6 months (3 months in the GC grup, 3 months in the GFA one).

ELIGIBILITY:
Inclusion Criteria:

* Clinical stable moderate to severe COPD (FEV1 <70%, FEV 1 / FVC <70%) total lung capacity (TLC> 80%) without conventional criteria for LTOT, optimal medical therapy, mean SpO2 ≤ 88% during the 6 minuts walking test and active life outside the home, other than active smoking or are in program respiratory rehabilitation.

Exclusion Criteria:

* Current smokers - Presence of respiratory failure and criteria for LTOT (PO2 <55 mmHg or 55-60 mmHg associated with pulmonary arterial hypertension, chronic cor pulmonale, congestive heart failure, arrhythmias or polycythemia). - Presence of impaired mobility - Cognitive impairment or intellectual disability to fill in questionnaires - No acceptance of liquid oxygen - Presence of active comorbidities (cardiovascular disease, rheumatologic, renal, hepatic) - Participation in pulmonary rehabilitation programs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2015-09; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Benefits on HRQOL | 3 months
  The aim is to analyze the benefits on HRQOL of suitable correction of desaturation in COPD patients without conventional criteria for OCD but with exercise desaturation.

SECONDARY OUTCOMES:
Reduce breathlessness during exercise | 3 months
  Reduce breathlessness during exercise
Increase exercise capacity | 3 months
  Increase exercise capacity
Increasing physical activity | 3 months
  Increasing physical activity

CONTACTS AND LOCATIONS:
Overall Officials: JULIA TARREGA, PhD, Principal Investigator — Hospital General de Granollers
Locations (1):
- Hospital General de Granollers, Granollers, BArcelona, Spain

REFERENCES:
- [Background] Continuous or nocturnal oxygen therapy in hypoxemic chronic obstructive lung disease: a clinical trial. Nocturnal Oxygen Therapy Trial Group. Ann Intern Med. 1980 Sep;93(3):391-8. doi: 10.7326/0003-4819-93-3-391. PMID 6776858
- [Background] Long term domiciliary oxygen therapy in chronic hypoxic cor pulmonale complicating chronic bronchitis and emphysema. Report of the Medical Research Council Working Party. Lancet. 1981 Mar 28;1(8222):681-6. PMID 6110912
- [Background] Andersson A, Strom K, Brodin H, Alton M, Boman G, Jakobsson P, Lindberg A, Uddenfeldt M, Walter H, Levin LA. Domiciliary liquid oxygen versus concentrator treatment in chronic hypoxaemia: a cost-utility analysis. Eur Respir J. 1998 Dec;12(6):1284-9. doi: 10.1183/09031936.98.12061284. PMID 9877478
- [Background] Bradley JM, Lasserson T, Elborn S, Macmahon J, O'neill B. A systematic review of randomized controlled trials examining the short-term benefit of ambulatory oxygen in COPD. Chest. 2007 Jan;131(1):278-85. doi: 10.1378/chest.06-0180. PMID 17218587
- [Background] Jolly EC, Di Boscio V, Aguirre L, Luna CM, Berensztein S, Gene RJ. Effects of supplemental oxygen during activity in patients with advanced COPD without severe resting hypoxemia. Chest. 2001 Aug;120(2):437-43. doi: 10.1378/chest.120.2.437. PMID 11502641
- [Background] Nonoyama ML, Brooks D, Guyatt GH, Goldstein RS. Effect of oxygen on health quality of life in patients with chronic obstructive pulmonary disease with transient exertional hypoxemia. Am J Respir Crit Care Med. 2007 Aug 15;176(4):343-9. doi: 10.1164/rccm.200702-308OC. Epub 2007 Apr 19. PMID 17446339